CLINICAL TRIAL: NCT06948318
Title: A Phase 3, Open-label, Multicenter Continuation Trial to Evaluate the Long-term Safety and Efficacy of Mezagitamab Subcutaneous Injection in Adults With Chronic Primary Immune Thrombocytopenia
Brief Title: A Continuation Study of Mezagitamab in Adults With Chronic Primary Immune Thrombocytopenia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-079-3003; 2025-521692-31-00 (EU CTIS Number)
Record Dates: First submitted 2025-04-25; First posted 2025-04-29 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Immune Thrombocytopenic Purpura (ITP)
Keywords: TAK-079; Immune Thrombocytopenia; Chronic Primary Immune Thrombocytopenia; Blood Platelet Disorders; Hematologic Diseases; Cytopenia; Purpura; Hemorrhagic Disorders; Autoimmune Diseases; Immune System Diseases; Hemorrhage; Skin Manifestations; Purpura, Thrombocytopenic, Idiopathic; Purpura, Thrombocytopenic
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Blood Platelet Disorders; Hematologic Diseases; Cytopenia; Purpura; Hemorrhagic Disorders; Autoimmune Diseases; Immune System Diseases; Hemorrhage; Skin Manifestations; Purpura, Thrombocytopenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mezagitamab (Experimental): Eligible participants who completed the TAK-079-3002 or TAK-079-1004 studies can receive on-demand treatment in this continuation study. The on-demand treatment course may be repeated as needed based on the pre-specified on-demand dosing criteria and investigator's clinical judgement.
  Interventions: Drug: Mezagitamab

INTERVENTIONS:
Drug: Mezagitamab — Mezagitamab injection administered SC.
  Other Names: TAK-079

SUMMARY:
Primary immune thrombocytopenia (ITP) is a condition where the immune system mistakenly destroys platelets, which are cells that help stop bleeding. This leads to a lower number of platelets, making it easier to bruise or bleed. The main aim of this study is to check how safe mezagitamab is and how well it is tolerated by adults with chronic primary ITP, if given over a longer time. Other aims are to learn how effective treatment with mezagitamab is and how the body processes it (called pharmacokinetics or PK) over a longer time.

Participants of the following previous mezagitamab studies will be invited to join this continuation study: TAK-079-3002 and TAK-079-1004. In this continuation study, participants will receive mezagitamab when certain protocol criteria are met.

During the study, participants will visit their study clinic several times.

ELIGIBILITY:
* Key Inclusion Criteria:

  1. The participant has completed TAK-079-3002 (end of trial [EOT]) or TAK-079-1004 (EOT).
* Key Exclusion criteria:

For TAK-079-3002 participants:

1. The participant has a history of severe allergic or anaphylactic reactions to recombinant proteins or excipients used in the mezagitamab formulation.

For TAK-079-1004 participants:

1. The participant has had any thrombotic or embolic event within 12 months before signing the ICF.
2. The participant has had a splenectomy within 3 months before signing the ICF.
3. The participant has active infection with hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV).
4. History of malignancy (including myelodysplastic syndrome) within 5 years of signing the ICF, except for treated non-melanoma skin cancer or cervical carcinoma in situ.
5. In the opinion of the investigator, the participant has a serious medical or psychiatric illness that could potentially interfere with the completion of treatment according to this protocol.
6. The participant has received anti-cluster of differentiation (CD) 20 treatment within 12 months before screening and either of the following applies:

   1. The last dose was received within 6 months before screening.
   2. The last dose was received between 6 and 12 months before screening and the participant has a CD19+ count below the lower limit of normal.
7. The participant has received any monoclonal or polyclonal antibody for immunomodulation within 6 months before Visit 1.
8. The participant has been exposed to another investigational agent within 4 weeks or 5 half-lives, whichever is longer, before Visit 1.
9. The participant has used anticoagulants (for example, vitamin K antagonists, direct oral anticoagulants) within 3 weeks prior to Visit 1.

10 The participant has received a live or live-attenuated vaccine within 4 weeks prior to the first dose of trial treatment or has any live or live-attenuated vaccine planned during the trial.

11. The participant has used the following immunosuppressive agents as specified prior to Visit 1: alkylating agents (for example, cyclophosphamide) within 8 weeks, vinca alkaloids (for example, vincristine) within 4 weeks, sulfones (for example, dapsone) within 3 weeks, antiproliferative agents: (for example, mycophenolate mofetil and azathioprine) within 2 weeks, and calcineurin inhibitors: (for example, cyclosporine) within 2 weeks.

12. The participant has a history of severe allergic or anaphylactic reactions to recombinant proteins or excipients used in the mezagitamab formulation.

Other protocol defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2029-07-29 (Estimated); Study Completion 2029-07-29 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious TEAEs | Up to approximately 108 weeks
  An adverse event (AE) is any untoward medical occurrence in a clinical trial participant, temporally associated with the use of the trial intervention, whether or not the occurrence is considered related to the trial intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of the trial intervention. TEAEs are defined as AEs with start dates at the time of or following the first exposure to mezagitamab in the parent trial for Cohort 1 and in this trial for Cohort 2. A serious TEAE is a TEAE that meets 1 or more of the criteria: results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or was otherwise considered medically important.
Number of Participants With TEAEs Leading to Permanent Withdrawal of Mezagitamab | Up to approximately 108 weeks
  An AE is any untoward medical occurrence in a clinical trial participant, temporally associated with the use of the trial intervention, whether or not the occurrence is considered related to the trial intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of the trial intervention. TEAEs are defined as AEs with start dates at the time of or following the first exposure to mezagitamab in the parent trial for Cohort 1 and in this trial for Cohort 2.

SECONDARY OUTCOMES:
Duration of Platelet Response | Up to approximately 108 weeks
  The duration of platelet response will be measured by the cumulative number of weeks on which platelet count was ≥30,000/microliters (μL) and ≥50,000/μL throughout the trial.
Duration Between On-Demand Treatment Courses | Up to approximately 108 weeks
Time to Initiation of the First On-Demand Treatment Course | Up to approximately 108 weeks
Number of Participants With Complete Response | Up to approximately 108 weeks
  Complete response is defined as achieving platelet counts ≥100,000/μL on at least 2 visits.
Number of Participants With Immune Thrombocytopenia (ITP) Remission | Up to approximately 108 weeks
  ITP Remission is defined as all platelet counts ≥50,000/μL for at least 24 weeks after any mezagitamab treatment cycle in the absence of further therapy for ITP.
Number of Participants With Reduction in Dose and/or Frequency of Concomitant ITP Medications | Up to approximately 108 weeks
  Concomitant ITP medications are defined as those given in addition to the trial intervention to treat your ITP. These medications include corticosteroids, thrombopoietin receptor agonists (TPO-RA), or fostamatinib.
Number of Participants Requiring Rescue Therapy | Up to approximately 108 weeks
Serum Concentrations of Mezagitamab | Pre-dose and at multiple time points post-dose up to Week 104
Number of Participants With Anti-Drug Antibodies (ADA) | Pre-dose and at multiple time points post-dose up to Week 104
Number of Participants With Neutralizing Antibody (NAb) | Pre-dose and at multiple time points post-dose up to Week 104

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (97):
- United States (17):
  - USC Norris Comprehensive Cancer Center - Keck Medicine of USC, Los Angeles, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Georgetown University Medical Center - Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - The University of Iowa, Iowa City, Iowa
  - University Of Louisville Brown Cancer Center, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Massachusetts Chan Medical School, Worcester, Massachusetts
  - Duke University Hospital, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - Perelman Center for Advanced Medicine (PCAM) Hospital of The University of Pennsylvania Penn Blood Disorders Program, Philadelphia, Pennsylvania
  - Lewis Katz School of Medicine at Temple University, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - University of Washingto, Seattle, Washington
  - Versiti Wisconsin, Inc, Milwaukee, Wisconsin
- Australia (10):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Concord Repatriation General Hospital, Concord, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - University of New South Wales (UNSW) - Liverpool Hospital - Liverpool Cancer Therapy Centre, Liverpool, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Monash University - Australian Centre for Blood Diseases (ACBD), Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Perth Blood Institute, West Perth, Western Australia
- Bulgaria (5):
  - Military Medical Academy Multiprofile Hospital for Active Treatment - Sofia, Sofia, Sofia-Grad
  - Medical Center "Fama Medical", Plovdiv
  - UMHAT Sv. Ivan Rilski, Sofia
  - UMHAT SofiaMed, OOD, Sofia
  - University Multiprofile Hospital for Active Treatment - Prof. Dr. Stoyan Kirkovich AD, Stara Zagora
- China (16):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hebei
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Soochow University - Shizijie Campus, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University - Donghu Campus, Nanchang, Jiangxi
  - Shengjing Hospital of China Medical University - Nanhu Campus, Shenyang, Liaoning
  - Shaanxi Provincial People's Hospital, Xi'an, Shaanxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Jinshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - Institute of Hematology and Blood Diseases Hospital Chinese Academy of Medical Sciences - PPDS, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Zhejiang Provincial Hospital of Chinese Medicine - Main, Hangzhou, Zhejiang
- Clinical Hospital Centar Zagreb, Zagreb, Croatia
- Queen Mary Hospital, Hong Kong, Pok Fu Lam, Hong Kong
- Azienda sanitaria universitaria Giuliano Isontina, Trieste, Italy
- Japan (13):
  - Chiba Aoba Municipal Hospital, Chuo-ku, Chiba
  - Chibaken Saiseikai Narashino Hospital, Narashino-shi, Chiba
  - National Hospital Organization Mito Medical Center, Ibaraki, Higashiibaraki
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Tohoku University Hospital, Sendai, Miyagi
  - Kansai Medical University Hospital, Hirakata-shi, Osaka
  - Hematology Ohta Clinic,Shinsaibashi, Osaka, Osaka
  - Osaka University Hospital, Suita-shi, Osaka
  - Saitama Medical University Hospital, Iruma-gun, Saitama
  - The University of Tokyo Hospital, Bunkyo-ku, Tokyo
  - Nihon University Itabashi Hospital, Itabashi-ku, Tokyo
  - Tokyo Metropolitan Bokutoh Hospital, Sumida-ku, Tokyo
  - Yamanashi Prefectural Central Hospital, Kofu, Yamanashi
- Netherlands (2):
  - Erasmus Medical Center, Department of Hematology, Rotterdam, South Holland
  - Hagaziekenhuis, The Hague, South Holland
- Poland (4):
  - IN-VIVO sp. z o.o., Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Instytut Hematologii i Transfuzjologii Klinika Zaburzen Hemostazy i Chorob Wewnetrznych, Warsaw, Masovian Voivodeship
  - Pratia Onkologia Katowice - PRATIA, Katowice, Silesian Voivodeship
  - N. Copernicus Provincial MCOT in Lodz, Lodz, Łódź Voivodeship
- South Korea (7):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Kyungpook National University Hospital, Daegu
  - Seoul National University Hospital (SNUH), Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Asan Medical Center, Seoul
- Spain (5):
  - Hospital Universitario Fundacion Alcorcon, Alcorcón, Mardrid
  - Hospital General Universitario Gregorio Maranon, Madrid, Mardrid
  - Hospital Universitario 12 de Octubre, Madrid, Mardrid
  - Hospital Universitario De Salaman, Salamanca
  - Hospital Universitario Virgen del Rocio, Seville
- Turkey (Türkiye) (5):
  - Ankara University Faculty of Medicine Cebeci Hospital, Department of Hematology, Mamak, Ankara
  - Aydin Adnan Menderes University Medical Faculty-Hematology Department, Efeler, Aydın
  - Cerrahpasa Tip Fakultesi, Edirne
  - Trakya Universitesi Tip Fakultesi Hastanesi, Edirne
  - Sakarya University Education and Research Hospital, Sakarya
- United Kingdom (10):
  - University Hospitals of Leicester NHS Trust, Leicester, East Midlands
  - Southampton General Hospital, Southampton, Hampshire
  - Guy's Hospital - Guy's & St. Thomas NHS Foundation Trust, Southwark, London
  - Royal Liverpool and Broadgreen University Hospitals NHS Trust, Liverpool, Merseyside
  - Greater Glasgow Health Board, Glasgow, Scotland
  - University Hospitals of North Midlands NHS Trust, Royal Stoke University Hospital, Stoke-on-Trent, Staffordshire
  - Leeds Teaching Hospitals NHS Trust, Leeds, Yorkshire
  - Barts Health NHS Trust, Royal London Hospital, London
  - University College London Hospitals, London
  - Imperial College Healthcare NHS Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/a3da95a29a994831??page=1&idFilter=TAK-079-3003